CLINICAL TRIAL: NCT04020458
Title: Dental Intervention Plan for Chronic Kidney Disease Patients Awaiting or With Kidney Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding lapse and poor enrollment rate
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Christopher Cutler, Chair and Professor, Augusta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1295706
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease; Chronic Periodontitis, Generalized, Moderate
Keywords: Kidney transplant, Immunoprofiling
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Periodontitis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontitis, no kidney disease (Active Comparator): Dental intervention i. Full mouth intraoral X-rays (FMX)
  ii. Full periodontal exam, diagnosis, Oral hygiene instructions (OHI)
  iii. RX: 7 days of p.o. metronidazole (250mg)/amoxicillin (500mg) T.I.D., combined with local chlorhexidine rinses (not for subjects with Kidney transplant).
  iv. Single visit intensive scaling and root planning (SRP) (full mouth)
  v. Re-evaluation after 4-6 weeks (referral for definitive treatment)
  vi. Extraction of teeth deemed hopeless based on periodontal, endodontic or restorative considerations
  vii. Caries control, sedative dressing (palliative), referral to endodontic dentist for root canal treatment (RCT)
  Interventions: Procedure: dental intervention
- Experimental- chronic kidney disease (Active Comparator): Dental intervention i. Full mouth intraoral X-rays (FMX)
  ii. Full periodontal exam, diagnosis, Oral hygiene instructions (OHI)
  iii. RX: 7 days of p.o. metronidazole (250mg)/amoxicillin (500mg) T.I.D., combined with local chlorhexidine rinses (not for subjects with Kidney transplant).
  iv. Single visit intensive scaling and root planning (SRP) (full mouth)
  v. Re-evaluation after 4-6 weeks (referral for definitive treatment)
  vi. Extraction of teeth deemed hopeless based on periodontal, endodontic or restorative considerations
  vii. Caries control, sedative dressing (palliative), referral to endodontic dentist for root canal treatment (RCT)
  Interventions: Procedure: dental intervention
- Control- no Periodontitis or kidney disease. (No Intervention): Only regular dental cleaning

INTERVENTIONS:
Procedure: dental intervention — Dental intervention plan for Group 1 and 3 subjects with periodontitis only, i) Full mouth intraoral X-rays (FMX)
  ii. Full periodontal exam, diagnosis, Oral hygiene instructions (OHI)
  iii. RX: 7 days of p.o. metronidazole (250mg)/amoxicillin (500mg) T.I.D., combined with local chlorhexidine rinses (not for subjects with Kidney transplant).
  iv. Single visit intensive scaling and root planning (SRP) (full mouth)
  v. Re-evaluation after 4-6 weeks (referral for definitive treatment)
  vi. Extraction of teeth deemed hopeless based on periodontal, endodontic or restorative considerations
  vii. Caries control, sedative dressing (palliative), referral to endodontic dentist for root canal treatment (RCT)
  Arms: Experimental- chronic kidney disease; Periodontitis, no kidney disease

SUMMARY:
The study aims to understand why dental infections in end-stage kidney patients results in poor outcomes for kidney functions and eventually transplant. Further, if an active dental treatment is provided to such patients, does it helps improve the kidney functional parameters, and eventually results in better survival of kidney transplant. In addition, the molecular markers that result in altered interactions between the blood cells and bacteria in these patients will be identified and compared with those found in a healthy subjects, or subjects with gum disease but no kidney disease. Besides, if any of the makers of altered interactions found in the blood can be found to be altered in the saliva samples from the patients with gum disease (periodontitis), and kidney disease, it will help to develop a non-invasive oral risk test for predicting outcomes of kidney transplant survival.

DETAILED DESCRIPTION:
PURPOSE: The Dental College of Georgia (DCG) and the Periodontics and Oral Health and Diagnostic Sciences departments propose to develop a collaborative clinical and research program with the Carlos and Marguerite Mason Trust Solid Organ Transplant Center at the Augusta University (AU) Medical Center. The overall goal is to develop a dental intervention program, with a research component, to address the role of dental infections in kidney transplantation outcomes, with the goal of improving best practices for kidney transplant patients. The study, which has been funded by the Mason Trust (C.W. Cutler, PI) is aimed toward improving overall quality of life of the patients on dialysis or with kidney transplant and reducing transplantation complications and failure rates.

AIM 1: To evaluate the effect of dental intervention on kidney transplant outcomes for patients with chronic kidney diseases awaiting kidney transplant/ or having received a kidney transplant within two (2) years. This aim will examine whether dental intervention will improve outcomes of patients with periodontitis (PD) and kidney disease, including kidney function and allograft survival in patients with chronic kidney diseases post-transplantation. Hypothesis is that active dental intervention will result in better oral health in patients with chronic kidney diseases resulting in better transplantation outcomes.

AIM 2: To determine the pathophysiological links between PD and chronic kidney disease with or without kidney transplantation.

Hypothesis is that active treatment of PD in chronic kidney patients will shift the systemic molecular profile towards anti-inflammatory, resulting in better transplant outcomes for these patients. The correlation of expression of various molecular proteins in saliva and blood will help to develop a non-invasive oral risk test for predicting outcomes of kidney transplant survival.

There will be three groups in the study:

Control groups: There will be 2 control groups. The data from these two groups will help establish the baseline for the different parameters to study in the experimental population.

1. Group 1: moderate to severe generalized periodontitis (PD) (no kidney disease).
2. Group 2: healthy controls, no PD or kidney disease.

Experimental group:

3) Group 3: Patients with chronic kidney disease : i. Group 3a- stage 5 (without dialysis, glomerular filtration rate (GFR) < 20)/ stage 5D (on dialysis), awaiting kidney transplant. (n=50) ii. Group 3b- Stages 2-4 (patients who have had either a living donor transplant (n=25), or deceased donor transplant within the last 2 years (n=25), with /without no history of rejection of kidney transplant) (total n=50).

The Group 1 and Group 2 subjects will be recruited from the patient population at AU-Dental College of Georgia (DCG), post-graduate periodontics clinic and/or primary care clinics at AU-Medical College of Georgia or volunteers who are willing to participate in this research study, after looking at study advertisements placed on DCG monitors or AU clinics. The group 3 patients will be recruited from among the patients registered at the AU Heath Kidney Transplant Center, who are either awaiting kidney transplant (Group 3a) or have received kidney transplant within last 2 years (Group 3b). The medical records of the potential will be reviewed against pre-screening criteria to determine their eligibility for the study. The eligible subjects will be invited for participating in the study.

At the pre-screening visit (visit 1), potential subjects will receive the Informed Consent Document (ICD) describing the overall aim of the study, study design, participation, and eligibility criteria. The consent process will occur in a separate room with no time restrictions. All questions and concerns will be clarified by the PI /Periodontics residents on the study or research coordinator. Consenting subjects will sign and date the consent form, and will receive a copy of the ICD. Any study procedure will be initiated only after obtaining a written, signed consent document from the potential subject. The consent document will be stored in a locked drawer in the research coordinators office at the Clinical Research Center, along with the subjects' records. At each of the subsequent visits (visits 2-8), eligible subjects will confirm consent to participate in the study.

Study procedures considered standard of care for all subjects:

1. Filling out a medical and dental history form
2. Being clinically examined by a dentist
3. Receiving oral hygiene instructions, oral health counseling, and referral for dental treatment
4. Dental intervention plan for Group 1 and 3 subjects with periodontitis only, considered standard of care i. Full mouth intraoral X-rays (FMX)

ii. Full periodontal exam, diagnosis, Oral hygiene instructions (OHI)

iii. RX: 7 days of p.o. metronidazole (250mg)/amoxicillin (500mg) T.I.D., combined with local chlorhexidine rinses (not for subjects with Kidney transplant).

iv. Single visit intensive scaling and root planning (SRP) (full mouth)

v. Re-evaluation after 4-6 weeks (referral for definitive treatment)

vi. Extraction of teeth deemed hopeless based on periodontal, endodontic or restorative considerations

vii. Caries control, sedative dressing (palliative), referral to endodontic dentist for root canal treatment (RCT)

Assessment of kidney function parameters, such as creatinine level and glomerular filtration rate, will be done at the AU Health Kidney Transplant Center for Group 3 subjects, as part of standard of care and follow-up visits at the clinic.

Study procedures for research purposes only on all subjects:

1. Phlebotomy for peripheral blood samples (15 mls per visit)
2. Sampling of dental plaque for microbiological analysis before and after dental intervention program (DIP)
3. Measurement of unstimulated and stimulated salivary flow rate measurement and
4. Collection of whole saliva for microbiological analysis, cytokine profile and other molecular markers.

Potential risks to subjects include

1. There is a small risk that subjects using antibiotics may have gastrointestinal problems.
2. There is a small risk that the use of mouth rinses can temporarily stain teeth light brown.
3. There is a small risk that the collection of a blood sample may cause major pain and bruising where the needle enters the skin, fainting and/or infection
4. There is a very small risk that periodontal probing, subgingival plaque sample collection, and dental anesthesia injections will cause major discomfort
5. There is a small risk that SRP may also cause major discomfort and pain
6. Withdrawal of fifteen (15) ml of blood from Group 3 subjects might put them at risk for anemia. Group 3 patients will be monitored at the AU-Health Kidney Transplant Clinic for anemia using CBC, hemoglobin and hematocrit levels.

Participants will be actively assessed for the occurrence of serious (SAEs) and non-serious adverse events (NSAEs) throughout the study. SAEs are defined as fatal or life-threatening events that require inpatient hospitalization or cause persistent or significant disability or incapacity. NSAEs are defined as any unfavorable and unintended sign, symptom, condition or disease temporally associated with a study intervention or medication. SAEs should be a rare occurrence and NSAEs are likely related but not restricted to procedures for biological sampling, scaling and root planning and antibiotic use including: inter-current illness, fever, nausea, vomiting, diarrhea, rashes, drug interactions, drug hypersensitivity, gingival pain, dentine hypersensitivity. Participants will be asked about any abnormal signs and symptoms and intra-oral examinations will be performed at every dental visit. Moreover, a phone number will be provided to participants for reporting any unexpected AE. Any occurrences will be recorded in preset forms and the following items will be assessed: description of the adverse event, period, frequency, severity, relationship with study procedures and medications, action taken and resolution. All SAEs will be reported to the IRB accordingly.

Confidentiality will be maintained by restricting access to subjects' data and de-identification of datasets and specimens. De-identification of the research records will be achieved by generating a subject study number. A separate list matching the subjects' study numbers and dental records will be kept in a separate file, which will be stored in a looked drawer in the research coordinator's office at the Clinical Research Center. Research team members will only have access to confidential data as needed for the strict execution of their functions. Subjects will not be identified by name in any report or publications resulting from this study.

For the purpose of statistical analysis, there will be 4 groups with experimental group 3a and 3b treated as separate groups.

As a preliminary step, the Shapiro-Wilk test will be used to assess normality of each dependent variable (DV). If the DV appears to be normally distributed, four-group repeated measures analysis based on a mixed effects regression model (MRM) will be performed. For each DV, MRMs will be used to assess the significance of each of the following design factors and covariates: (1) Within-subjects (repeated-measures) Factor: Time (6 levels: Baseline, 4 weeks, 3 months, 6 months, 1 year, 5 years); (2) Between-subjects Factor: Group (4 levels: Groups 1, 2, 3a, 3b); (3) Interaction terms: Time by Group, Group by selected covariates, Time by selected covariates; and (4) Covariates (age, race, sex, etc.). For each DV, several competing covariance structures for the repeated measures will be examined, including unstructured, compound symmetry, Huynh-Feldt, first-order autoregressive, first-order autoregressive with heterogeneous variances, etc. The Akaike (AIC) and Bayesian (BIC) Information Criteria will be used to select the most appropriate covariance structure. Tukey-Kramer adjustments will be made to any post-hoc multiple comparisons in order to control the family-wise error rate at the 0.05 level. If a DV appears to be non-normally distributed, an attempt will be made to identify a transformation to normality using the Box-Cox method. If an appropriate transformation cannot be found, robust multivariate analyses will be used instead of standard normal-theory based methods. All statistical analyses will be carried out using SAS 9.4, and all statistical tests will be performed using a two-tailed significance level of 0.05 unless otherwise specified.

ELIGIBILITY:
Inclusion and Exclusion Criteria

Inclusion and Exclusion Criteria List the inclusion/exclusion criteria:

There will be three groups in the study:

Control groups: There will be 2 control groups. The data from these two groups will help establish the baseline for the different parameters to be evaluated in the experimental population.

1) Group 1: moderate to severe generalized periodontitis (PD) (no kidney disease).

2) Group 2: healthy controls, no PD or kidney disease. Inclusion Criteria

1. Subjects of both sexes, 21 to 75 years of age will be included.
2. Subjects must have moderate to severe generalized periodontitis (PD) (Group 1) (n=50) or no PD (Group 2) (n=50). PD is defined as a patient in the 3rd or later decades of life with the presence of at least 20 natural teeth, >30% of which exhibit: probing depth > 6mm, attachment loss > 3 mm, bleeding on probing, alveolar bone crest > 3 mm from cemento-enamel junction [CEJ]. Healthy controls will also have > 20 teeth, but no alveolar bone loss, attachment loss or BOP and alveolar bone crest 1-2 mm from the CEJ.
3. No kidney disease
4. All potential subjects must sign an informed consent prior to study enrollment.

Exclusion Criteria

1. Periodontal treatment (i.e., surgical or nonsurgical) within 3 months prior to enrollment.
2. Treatment with antibiotics within 3 months prior to enrollment.
3. Presence of heart murmur, history of rheumatic fever, valvular disease, prosthetic joint replacement necessitating antibiotic prophylaxis.
4. Kidney disease
5. Cancer or chronic viral infections such as HIV and hepatitis B
6. Inability to take Metronidazole and Amoxicillin combination due to allergy.

Experimental group:

3) Group 3: Patients with chronic kidney disease : i. Group 3a- stage 5 (without dialysis, glomerular filtration rate (GFR) < 20)/ stage 5D (on dialysis), awaiting kidney transplant. (n=50) ii. Group 3b- Stages 2-4 (patients who have had either a living donor transplant (n=25), or deceased donor transplant within the last 2 years (n=25), with /without no history of rejection of kidney transplant) (total n=50).

Inclusion Criteria

1. Subjects of both sexes, 21 to 75 years of age will be included.
2. All potential subjects must sign an informed consent prior to study enrollment.
3. All potential subjects should be able to drive or be driven to the DCG for dental treatment and follow-up visits.
4. For Group 3b subjects, post-transplant group, glomerular filtration rate with creatinine clearance rate should be in the range of 1.5 - 1.9 ml/min. This will yield a more uniform subject population for statistical analysis of the data.

Exclusion Criteria

1. Active, chronic viral infections such as HIV, Hepatitis B, Hepatitis C (these patients are immunocompromised and on antiviral drugs, which might result in an altered immune profile for such patients).
2. Inability to take Metronidazole and Amoxicillin combination due to allergy or poor kidney function.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Kidney transplant outcome | 3 years
  % allograft survival

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Cutler, Principal Investigator — Dental College of Georgia-Augusta University
Locations (1):
- Augusta University-Dental College of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The data generate will be published and made available to anyone who requests for samples or data.